CLINICAL TRIAL: NCT06019429
Title: A Non-randomized Trial Testing the Efficiency of a Universal School-based Intervention Promoting Social-emotional Development and Self-esteem in Primary School Students
Brief Title: Promoting Social-emotional Development and Self-esteem in Primary School Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiteit Leiden (Other)
Responsible Party: Principal Investigator, Bianca Boyer, Assistant professor, Universiteit Leiden
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 158765324
Record Dates: First submitted 2023-08-01; First posted 2023-08-31 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Prosocial Behavior; Anxiety Disorders and Symptoms; Attention Deficit Hyperactivity Disorder; Healthy; Emotional Problem; Self Esteem; Peer Group
Keywords: prosocial behavior; anxiety; self esteem; classroom peer context; attention deficit hyperactivity disorder
MeSH Terms: conditions — Altruism; Anxiety Disorders; Attention Deficit Disorder with Hyperactivity | interventions — Schools

STUDY DESIGN:
Intervention Model Description: Schools who partake in this study decide the type of program they will receive: HiRO without judo, HiRO with judo, school-as-usual
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HiRO plus judo (Experimental): In this condition, students receive weekly classes aimed to promote social-emotional development. In addition, they will receive 6 judo classes.
  Interventions: Behavioral: HiRO +judo
- HiRO (Experimental): In this condition, students receive weekly classes aimed to promote social-emotional development.
  Interventions: Behavioral: HiRO
- School as usual (Active Comparator): In this condition, students receive any amount of classes organized by their school to promote social-emotional development.
  Interventions: Behavioral: School as usual

INTERVENTIONS:
Behavioral: HiRO — HiRO consists of weekly lessons. The lessons are aimed to promote social-emotional development. More specifically, lessons are designed to develop and enhance 1) trust, 2) collaboration, 3) respect, 4) self control, 5) resilience, 6) discipline, 7) joy. The annual program consists of four phases:
  Phase 1 & 3: Fundamental phase (6 weeks) Engaging with the values through movement. In these phases, group formation and establishing behavioral expectations are central. In the Fundamental phase, one value is addressed school-wide each week. The entire school starts with trust and ends with discipline.
  Phase 2 & 4: Theme weeks (12 lessons) A customized series of Experiential lessons for each class. Experiential learning is the guiding principle of the program, with a strong foundation based on the values upheld in judo. The learning cycle forms the basis for each experiential lesson within HiRO, and focusses on concrete experience, reflective observation, conceptualization, and practice.
  Arms: HiRO
Behavioral: HiRO +judo — In the condition HiRO with judo, students receive the same treatment as offered in the HiRO condition. In addition, they receive physical judo classes that are designed to translate the above-mentioned values to the behavioral level.
  Arms: HiRO plus judo
Behavioral: School as usual — Any amount of classes offered to promote social-emotional development
  Arms: School as usual

SUMMARY:
This is an effectiveness study into a program ("HiRO") for improving social-emotional development, self esteem and the perceived classroom peer context in primary school students (aged 4-13 years). To this end, schools are divided into three conditions based on the choice of the schools (non-randomized): 1) School As Usual, 2) HiRo without judo classes, and 3) HiRO with judo classes. In all participating schools, social-emotional skills, self-image, emotional problems, and classroom peer context are measured three times by means of questionnaires (both self-report and parent-report).

In The Netherlands primary schools are obliged to offer students training in social-emotional development. Schools can decide to develop their own program or make use of existing programs delivered by third parties, such as HiRO. In this study HiRO is compared to school as usual, that is, any other program offered to promote social -emotional development than HiRO.

The main questions to answer are:

* What is the effect of HiRO on the development of prosocial behavior?
* What is the effect of HiRO on the development of emotional problems (depression, anxiety)?
* What is the effect of HiRO on self-esteem?
* What is the effect of HiRO on perceived peer context?

Researchers will compare HiRO with and without judo to "school as usual" testing the following hypotheses:

HiRO will result in increased prosocial skills as compared to school as usual. HiRO will result in decreased emotional problems as compared to school as usual.

HiRO will result in increased self-esteem as compared to school as usual. HiRO will result in improved perceived peer context as compared to school as usual.

DETAILED DESCRIPTION:
This is a non-randomized trial, with a 3 (time) x 3 (condition) within-between subjects design.

All children (and their parents) within the participating primary schools are asked to join this study. Independent of participation in this study, all children in these schools will receive the intervention as it is part of the curriculum focussing on the development of prosocial skills.

Schools will be called to ask if participants would like to participate in the study: schools choose in what condition participation is desired. In march/april 2023: schools share information letter with parents by email/in school app with a link to the informed consent. In june 2023: during end-of-the-year meetings with parents, teachers will approach parents that have not responded yet whether participation is approved. In addition, children in group 8 (with possible children of 12 years and older) will get information from teachers about the study and an information letter. Subsequently, children will be asked whether participation is approved. Assessements will take place in classrooms of the participating schools during school hours for children 8 years and older. For children younger than 8 years parent report will be used.

This study will obtain a data set with a hierarchical structure. The three observations are nested within students, students are nested within classrooms and classrooms are nested within schools. Therefore, a three-level growth model will be used. Lee and Hong (2021) provided sample size guidelines based on simulation studies for three-level growth models using Monte Carlo methods while considering various realistic ICC values at the three levels. The conservative estimation is made that only 10 out of 23 (average number of students per class) students per class participate in this study. Therefore the simulation results of Lee and Hong (2021) provided for 10 students per group are considered. Across all fixed effects and an intraclass correlation coeffcient at level 3 (schools) of .15, 2 out of 6 power rates were found to be below the .80 level, when 50 groups are included. With 100 groups included, all power rates were found to exceed .87. Based on these numbers, the aim is to include 75 groups in total, bringing the total number of participating students (again assuming 10 participants per group) to 10x75 = 750.

Multilevel regression analyses will be performed to evaluate the effect of HiRO on social-emotional development, self-esteem, and the perceived classroom peer context. Multilevel analyses is an intent-to-treat procedure that does not impute missing data but deals with incomplete data by assuming that the available data for a given subject are representative of that subject's deviation from the average trends across time. The level1 model includes the time variable, which captures within-person variation over time, in the level 2 model between person characteristics such an intervention condition are used to predict the slope estimates. In the level 3 model between group characteristics can be modeled.

ELIGIBILITY:
Inclusion Criteria:

All primary school children

Exclusion Criteria:

None

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Prosocial behavior | Up to 11 months
  The Strengths and Difficulties Questionnaire (SDQ) is a self-report and third-party informant (parent and teacher) screening instrument for psychosocial functioning of children and adolescents (Goodman, 1997); Dutch version (Widenfelt, Goedhart, Treffers, & Goodman, 2003). For 8 to 13 year old participants, both the self-report and parent version is used. For 4-7 year old participants only the parent version is used. The SDQ is comprised of five subscales: (a) emotional symptoms, (b) conduct problems, (c) hyperactivity/ inattention, (d) peer relationship problems, and (e) prosocial behavior. All subscales consist of five items using a 3-point Likert scale (ranging from 0 = ''not true'' to 2 = ''very true'' The SDQ is a reliable and valid screener of psychological difficulties across social-emotional domains (Muris, Meesters, & Van den Berg, 2003; Van Rooy, Veenstra, Clench-Aas, 2008).

SECONDARY OUTCOMES:
Self-esteem | Up to 11 months
  The child version of the Rosenberg's Self Esteem Scale (CRSES; Wood, Griffin, Barton, Sandercock, 2021) has been developed to assess self esteem in children aged 7-12 years. The CRSES comprises five positive and five negative statements each with four possible responses scored from one to four. Scoring is reversed for responses to negative items so that a higher score indicates better overall self esteem. A validation study has tested the internal consistency, convergent validity, and factor structure of the CRSES. A unidimensional factor structure provided an adequate fit, and total scores were related to life satisfaction. As the sample also consists of children aged 4-7 years of age, a 10-item parent version of the Rosenberg Self Esteem Scale (RSES) was developed that will be validated using the pre-treatment assessment of this trial.

OTHER OUTCOMES:
Anxiety and emotional problems | Up to 11 months
  The Youth Anxiety Measure for the Diagnostic and Statistical Manual of Mental Disorders (YAM-5) is a self- and parent-report questionnaire to assess anxiety disorder symptoms in children and adolescents. Part one, used in this study, consists of 28 items and measures the 5 major anxiety disorders including separation anxiety disorder, selective mutism, social anxiety disorder, panic disorder, and generalized anxiety disorder. The five subscales consist of four to seven items using a 4-point Likert scale (ranging from 0 = ''never'' to 3 = 'always''. Higher scores indicate higher levels of anxiety. A validation study demonstrated that the measure was easy to complete by youngsters, support was found for the psychometric qualities of the measure: that is, the internal consistency was good for both parts, as well as for most of the subscales, the parent-child agreement appeared satisfactory, and there was also evidence for the validity of the scale.
Classroom Peer Context Questionnaire (CPCQ) | Up to 11 months
  The Classroom Peer Context Questionnaire (CPCQ) is a self-report questionnaire that can be used to assess the self-perceived peer context in the classroom. The questionnaire consists of 20 items belonging to 5 scales; comfort, cooperation, conflict, cohesion and isolation.Confirmatory factor analyses supports these 5 dimensions. Good reliability, validity, and stability for each dimension has been demonstrated.

CONTACTS AND LOCATIONS:
Overall Officials: Bianca Boyer, PhD, Principal Investigator — Leiden University
Locations (1):
- Leiden University, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No